CLINICAL TRIAL: NCT05273450
Title: Promoting Smoking Cessation Among Individuals With Food Insecurity: Promoting the Use of Evidence-Based Tobacco Cessation Resources Through Community Food Pantries
Brief Title: An Intervention to Promote Use of Smoking Cessation Resources Among Adults Using Community Food Pantries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Jin Kim-Mozeleski, Assistant Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Kim-MozeleskiStudy20211283
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Smoking Cessation; Food Insecurity
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quitline Information with Reinforcement (Experimental)
  Interventions: Behavioral: Quitline Information with Reinforcement
- Quitline Information Only (No Intervention)

INTERVENTIONS:
Behavioral: Quitline Information with Reinforcement — The intervention arm involves direct referral to the Ohio Tobacco Quitline, with up to two brief follow-up telephone calls from the research team to elicit motivation to quit, emphasize benefits of calling the quitline, encourage use and address concerns. Participants are surveyed at baseline and at 3-month follow-up to assess awareness and use of the quitline.
  Arms: Quitline Information with Reinforcement

SUMMARY:
The primary objective of this pilot randomized controlled study is to raise awareness and use of an evidence-based tobacco cessation resource that is underutilized among smokers (the Ohio Tobacco Quitline), specifically targeting Cleveland-area residents who have experiences with food insecurity. The study will assess the feasibility and acceptability of conducting informational outreach on tobacco cessation resources in community settings in which there is a relatively high proportion of tobacco users (i.e., food pantries). The study will derive preliminary estimates regarding the effectiveness of tobacco cessation outreach, by assessing whether outreach activities result in changes in awareness/knowledge of the quitline and use/engagement of the quitline.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 or older
* Current tobacco smoker willing to receive information about quitting resources
* Lives in Cuyahoga County, Ohio
* Has a reliable telephone number and an email address

Exclusion Criteria:

* Aged 20 or younger
* Current non-smoker, or current smoking who is not willing to receive information about quitting resources
* Lives outside Cuyahoga County, Ohio
* Does not have a reliable telephone number and an email address

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Awareness of the quitline | 3 months
  How familiar are you with the Ohio Tobacco Quitline? (a) Not familiar at all - I have not heard about the quitline, (b) Somewhat familiar - I have heard of the quit line but have not used it, (c) Familiar - I have used their services but it was over a year ago, (d) Very familiar - I am currently connected to their services
Use of the quitline | 3 months
  After enrolling in this research study [past 3 months], did you receive a referral to the Ohio Tobacco Quitline? (a) Yes, and I enrolled, (b) Yes, but I did not enroll, (c) No
Use of the quitline | 3 months
  In the past 3 months, which of the following methods did you try to stop smoking? 'Called the Ohio Tobacco Quitline' is checked

CONTACTS AND LOCATIONS:
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT05273450/ICF_000.pdf